CLINICAL TRIAL: NCT07335250
Title: Postoperative Pain Control With Intertransverse Process Block in Patients Undergoing Thoracotomy With Lobectomy
Brief Title: Intertransverse Process Block for Postoperative Analgesia After Thoracotomy and Lobectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Ömer Keklicek, principal investigator, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025/485
Record Dates: First submitted 2026-01-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Acute Postoperative Pain; Thoracotomy Surgery; Intertransverse Process Block
Keywords: Intertransverse Process Block; Thoracotomy Lobectomy; Acute Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two parallel groups to receive either an ultrasound-guided intertransverse process block with bupivacaine or a placebo saline injection at the same site. Each participant will receive only one intervention, and postoperative outcomes will be compared between the two groups.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The study is triple-blinded. Neither the participants, the block performer, nor the outcome assessors are aware of the group assignments. Randomization codes are stored centrally, and a separate staff member who is not involved in patient care or outcome assessment prepares the study solutions and labels them in an identical manner to maintain allocation concealment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block Group - Intertransverse Process Block (Active Comparator)
  Interventions: Procedure: Intertransverse Process Block
- Control Group - Placebo: (Placebo Comparator)
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Intertransverse Process Block — The block will be performed under ultrasound guidance by the same anesthesiologist with more than five years of experience, immediately after surgery and before emergence from anesthesia. Patients will be placed in the lateral decubitus position with the operative side uppermost and the skin prepared.
  Using a high-frequency linear probe (Mindray DC-60 Exp), the T5 spinous process will be identified at the midline, then the probe will be moved approximately 2 cm laterally to visualize the superior costotransverse ligament (SCTL) and pleura. The needle will be advanced in-plane in a caudal-to-cranial direction toward the cranial border of the fourth rib. After confirmation of correct spread by hydrodissection, 20 mL of 0.5% bupivacaine will be injected.
  Arms: Block Group - Intertransverse Process Block
Procedure: Placebo — In the control group, the same procedure will be conducted, but saline will be injected instead of local anesthetic.
  Arms: Control Group - Placebo:

SUMMARY:
This prospective, randomized, triple-blind, placebo-controlled clinical trial will investigate the effectiveness of the intertransverse process block (ITPB) for postoperative analgesia in patients undergoing elective thoracotomy with unilateral lobectomy. The study will be conducted at a single tertiary center in accordance with the principles of the Declaration of Helsinki, and written informed consent will be obtained from all participants.

Patients will be randomized in a 1:1 ratio to receive either ultrasound-guided ITPB with 0.5% bupivacaine or placebo (normal saline) prepared in identical syringes to ensure allocation concealment. The block will be performed by an experienced anesthesiologist immediately after surgery and before emergence from anesthesia. Both groups will receive standardized general anesthesia, multimodal perioperative analgesia, and postoperative intravenous morphine patient-controlled analgesia (PCA).

The trial aims to evaluate the analgesic efficacy and opioid-sparing effect of ITPB while maintaining safety and adherence to routine clinical practice. Outcomes will include postoperative pain scores, opioid consumption, rescue analgesia requirement, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent

Age between 18 and 85 years

ASA Physical Status classification I-III

Elective thoracotomy with planned unilateral lobectomy

Anticipated hospital stay of at least one night

Expected requirement for parenteral opioid analgesia for at least 24 hours postoperatively

Ability to operate an intravenous patient-controlled analgesia (PCA) device

Exclusion Criteria:

* Patients undergoing emergency surgery

Presence of infection or open wound at the injection site

Coagulopathy

Hepatic or renal failure

Patients undergoing reoperation

Patients with missing or incomplete data

Pregnancy or lactation

Tracheal malformation or tracheostomy

Chronic opioid use (≥30 days within the last 3 months, ≥15 mg/day morphine equivalent)

Patients exceeding the maximum safe local anesthetic dose based on weight (2.5 mg/kg, max 150 mg)

Patients who refuse data privacy consent will be excluded from the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Morphine Consumption Within the First 24 Hours After Surgery | 24 hours postoperatively
  The primary objective of the study is to evaluate the effect of the intertransverse process block (ITPB) on opioid consumption within the first 24 hours postoperatively in patients undergoing thoracotomy with unilateral lobectomy. Morphine consumption will be determined based on patient-controlled analgesia (PCA) use.

SECONDARY OUTCOMES:
NRS score | 0 to 24 hours postoperatively
  After extubation, patients will be assessed at 0, 6, 12, and 24 hours for pain intensity both at rest and during coughing using the Numeric Rating Scale (NRS; 0-10).
  The Numeric Rating Scale ranges from 0 (no pain) to 10 (worst pain imaginable), with higher scores indicating worse pain severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No